CLINICAL TRIAL: NCT02482558
Title: Investigating the Effects of a High GI Versus a Low GI Diet on Hepatic Metabolism and Satiety Levels in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UoN-URDC GI trial
Record Dates: First submitted 2015-01-30; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Glycaemic Index; NAFLD; Glycogen; Liver; Diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High GI diet (Experimental): 8 Healthy subjects will be assessed at the start and end of a 7 day high glycaemic in diet following the appropriate High/Low Glycaemic index test breakfast.
  Interventions: Other: High/Low Glycaemic index test breakfast
- Low GI diet (Experimental): 8 Healthy subjects will be assessed at the start and end of a 7 day low glycaemic in diet following the appropriate High/Low Glycaemic index test breakfast.
  Interventions: Other: High/Low Glycaemic index test breakfast

INTERVENTIONS:
Other: High/Low Glycaemic index test breakfast — High/Low Glycaemic index test breakfast on test days for a High/Low Glycaemic index 7-day diet

SUMMARY:
The aim of this study is to investigate the effect of a one week high versus low glycaemic index dietary intervention on hepatic glycogen and lipid levels and blood hormone levels in a two way cross overs study and to see if there is any correlation between this and satiety or appetite.

DETAILED DESCRIPTION:
8 Healthy subject will be scanned the start and end of a 7 day high versus low glycaemic in diet with a 4 week washout between arms. During scan days the hepatic glycogen response to a corresponding high versus low glycaemic index test meal will be measured using 13C Magnetic resonance spectroscopy (MRS) to explore any acute changes in metabolic response. Baseline liver lipid levels will be measured using 1H MRS to explore any long term changes in liver lipid levels.

Blood samples will also be obtained throughout the test day to measure for blood glucose, insulin and blood hormone response. Satiety surveys will also be taken throughout the test day and during the diet week.

The main hypothesis is that a one week calorie matched Glycaemic index varied diet will result in an altered response of liver glycogen levels acutely following a meal and also longer term hepatic liver lipid levels. A secondary hypothesis is that there will also be associated changes in blood sugar and hormone levels and that all these changes will have an effect on satiety levels in subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian
* Self-reported non-athletic but healthy: not carrying out strenuous exercise (no high sweat, out of breath, high heart rate activities and less than 2 hours moderate exercise a week), moderate drinkers (less than 3 units a day), no smokers
* Routinely eating 3 meals a day
* Stable weight
* Age ≥ 18 and ≤ 35
* Body mass index (BMI - weight / squared height ) ≥ 20.0 and ≤ 27.0 kg/m2
* Suitable for MRI scanning (e.g., absence of metal implants, infusion pumps and pacemakers) as assessed by the attached MRI safety questionnaire.
* Suitable for blood samples and cannula insertion (e.g., no aversion to needles)
* Willing to follow both prescribed diet plans
* Not taking any concurrent medication

Exclusion Criteria:

* No diabetics or other metabolic disorders (e.g. insulin resistance, thyroid dysfunction)
* No volunteers with liver disease
* No clotting disorders
* No Participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study.
* No use of any medically or self-prescribed diet from the moment of pre-study examination till the end of the study
* Taking prescription medication or any other drugs that may influence liver function or glucose and energy metabolism.
* Any allergy or food intolerance
* Unsuitable for MR scanning (i.e. have pacemakers and/or medical implants)
* The subject is an employee of Unilever or the site conducting the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Liver glycogen | 7 days
  Liver glycogen content was determined by Magnetic Resonance Spectroscopy using the distinct 13C signals from the glycogen polymer. The glycogen signal resonates at 101.4 ppm, and was calibrated using an external reference peak situated in the centre of the coil (175ppm) and quantified with reference to an ex vivo glycogen acquisition.

SECONDARY OUTCOMES:
Liver lipids | 7 days
  Liver lipid content was determined by Magnetic Resonance Spectroscopy using the distinct 1H signals from the fatty acid. The peak area of the main chain CH2 peak at 1.3ppm was calibrated using the water peak at 4.7ppm as an internal reference, corrected for T2 relaxation, and quantified using biological parameters.

OTHER OUTCOMES:
Blood glucose | 7 days
  Subjects were cannulated at the start of the test day by research nurses and samples taken regularly for blood glucose. Blood glucose levels were measured approximately every 20 minutes for the first 3 hours of the feeding trial, and then hourly after up to 5 hours. 0.1 ml samples were drawn into plastic fluoride/oxalate glucose preservation tubes and were assessed at the University of Nottingham.
Satiety ratings | 7 days
  During the experiment subjects filled out satiety questionnaires using Visual Analogue Scales (VAS) by answering each of five mixed appetite questions - "1. How hungry do you feel", "2. How satisfied do you feel", "3. How full do you feel?", "4. How strong is your desire to eat" and "5. How much do you think you can eat?". Subjects indicated their response by making a vertical mark on a horizontal scale between 1 and 10 every 20 minutes throughout the test day, and also before and after breakfast, lunch and dinner on days 1, 4 and 7 of the diet week.
Blood hormones | 7 days
  Subjects were cannulated at the start of the test day by research nurses and samples taken regularly for blood hormones. Blood hormone levels were measured every 20 minutes for the first 3 hours, and then hourly after up to 5 hours. 0.5 ml samples for analysis of hormone levels were drawn into Becton-Dickinson P800 tubes and were analyzed at Unilever R&D Colworth using multiplex assay kits from Millipore. The hormones assayed were Amylin, CCK, Ghrelin, Glucagon, GLP-1, GIP, Insulin, Leptin, PP and PYY.

CONTACTS AND LOCATIONS:
Overall Officials: Penny Gowland, PhD, Principal Investigator — School of Physics & Astronomy, University of Nottingham; Robin Spiller, MD, Principal Investigator — School of Medicine, University of Nottingham
Locations (1):
- Sir Peter Mansfield Magnetic Resonance Centre, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom